CLINICAL TRIAL: NCT04601883
Title: Colchicine Treatment for Patients With Hand Osteoarthritis: A Randomised, Placebo-controlled Trial.
Brief Title: Colchicine as Treatment for People With Hand Osteoarthritis
Acronym: COLOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henning Bliddal (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, MD, DMSci, Professor of Rheumatology, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APPI2-2020-AD03
Record Dates: First submitted 2020-10-12; First posted 2020-10-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis Hand; Osteoarthritis Finger
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Tablet colchicine 0.5 mg administered two times daily
  Interventions: Drug: Colchicine 0.5 MG
- Placebo (Placebo Comparator): Tablet placebo administered two times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — The intervention tablets are commercially available Colchicine "Tiofarma"
  Arms: Colchicine
Drug: Placebo — Encapsulated placebo tablets. Placebo is identical to the active intervention.
  Arms: Placebo

SUMMARY:
The study aims to compare oral colchicine 0.5 mg administered two times daily for 12 weeks with placebo as a treatment of hand OA symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Hand OA according to the ACR criteria above.
3. Hand OA finger pain: Pain at rest ≥40 mm on VAS (0 to 100 mm range).

Exclusion Criteria:

Comorbidities

1. Other known medical disease that may affect joints, e.g. RA, gout, PsA
2. Positive anti-cyclic citrullinated peptide (>10 kU/L)
3. Known cutaneous deposition diseases (e.g. amyloidosis or porphyria).
4. Known blood dyscrasias and coagulation disorders
5. Known malignancy (except successfully treated squamous or basal cell skin carcinoma)
6. Elevated alanine transaminase (>45 U/L females, >70 U/L for males)
7. Creatinine clearance ≤60 ml/min
8. Elevated creatine kinase (>210 U/L females, >280 U/L for males)
9. Known allergies towards the interventions
10. Drug or alcohol abuse in the last year
11. Generalised pain syndromes such as fibromyalgia
12. Current reflux
13. Current or recurrent diarrhoeal illnesses
14. Current abdominal pain
15. Known peripheral neuropathies
16. Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as e.g. psychiatric disorders.

    Medical history
17. History of hand surgery within 12 months prior enrolment.
18. History of arthroplasty or arthrodesis in the hand Management strategies
19. Treatment with P-glycoprotein inhibitors and/or cytochrome P450 3A4 (CYP3A4) inhibitors, see section "Colchicine safety in drug-drug interactions" and table 7. If potential participants have been treated with these pharmaceuticals previously, treatment must be terminated 5 half-lifes before initiation of study drug.
20. Use of systemic corticosteroids equivalent of ≥ 7.5 mg prednisolone daily within 3 months.
21. Participation in experimental device or experimental drug study 3 months prior to enrolment.
22. Intra-articular treatments or aspirations of any kind of any joint in the hands 3 months before inclusion
23. Intra-articular corticosteroids into any joint 1 months before inclusion
24. Current use of synthetic or non-synthetic opioids
25. Scheduled surgery during study participation
26. Planning to start other treatment for hand OA in the study participation period.

    Reproductive system
27. Pregnancy.
28. Planned pregnancy within the study period, 3 months after end of study treatment for female fertile participant and 6 months after end of study treatment for male participant.
29. Insufficient anti-conception therapy for female fertile participants within the study period and 3 months after end of study treatment. Sufficient anti-conception therapy consists of intra-uterine device (coil),hormonal anti-conception (birth control pills, implant, intra-uterine system, dermal patch, vaginal ring, or injections) or sexual abstinence Female participants are considered infertile if they are postmenopausal or if they have undergone surgical sterilisation (bilateral salpingectomy, hysterectomy or bilateral oophorectomy). Postmenopausal state is defined as no menses for 12 months without alternative medical cause before inclusion in the study. Menopause state will be confirmed by measurement of follicle stimulating hormone.
30. Insufficient anti-conception therapy for male participants within the study period and 6 months after end of study treatment. Sufficient anti-conception therapy consists of condom or sexual abstinence. Male participants are considered sterile if they have undergone surgical sterilisation (vasectomy).
31. Breast-feeding

A target hand will be selected for outcome assessment once individual fulfills in- and exclusions criterias. Selection of the target hand will adhere to the following, with advancement to next step if unable to choose target hand based on the given criteria.

1. The hand with most overall pain, assessed by VAS finger joint pain.
2. The hand with most overall reduced function, assessed by AUSCAN function subscale.
3. The hand with most overall stiffness, assessed by AUSCAN stiffness subscale.
4. The hand with most swollen joints, assessed by physician joint count.
5. The hand with most tender joints, assessed by physician joint count.
6. The hand with highest summed radiographic score, assessed by radiographic scoring of conventional X-ray.
7. If unable to select target hand based on the above criteria, a target hand will be randomly assigned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Finger pain | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, on changes in finger joint pain of the target hand from baseline to week 12, in patients with painful hand OA measured on a visual analogue scale spanning from 0 to 100, where 0 equals no symptoms and 100 equals worst imaginable symptoms.

SECONDARY OUTCOMES:
Function | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in function of both hands measured on the Australian/Canadian Hand Index Function Score spanning from 0 to 900, where higher scores equals worse function.
Thumb base pain | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in thumb base pain of the target hand measured on a visual analogue scale spanning from 0 to 100, where 0 equals no symptoms and 100 equals worst imaginable symptoms.
Pain hands | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in pain of both hands measured on the Australian/Canadian Hand Index Pain Score spanning from 0 to 500, where higher scores equals worse pain.
Joint activity | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in joint activity of the target hand measured on physician tender joint count
Patient global assessment | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in patient global assessment measured on a visual analogue scale spanning from 0 to 100, where 0 equals no symptoms and 100 equals worst imaginable symptoms.
Quality of life measured by European Quality of Life 5 Dimensions | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in quality of life measured on the European Quality of Life 5 Dimensions spanning from -0.624 to 1.000, where higher scores equals better quality of life.
Hand strength | Week 12
  To compare the effect of oral colchicine 0.5 mg bid, relative to placebo, from baseline to week 12, in patients with painful hand OA on changes in hand strength of the target hand measured on grippit
Number of treatment responders according to OMERACT-OARSI response criteria | Week 12
  The following two conditions is observed at the post-baseline assessment:
  1. In either pain (finger pain) or function (function), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 percent points (0-100 scale), OR
  2. Improvement in at least two of the following three:
     * Improvement in pain (finger pain) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale)
     * Improvement in function (function) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale)
     * Improvement in patient's global assessment defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dossing A, Henriksen M, Ellegaard K, Nielsen SM, Stamp LK, Muller FC, Kloppenburg M, Haugen IK, McCarthy GM, Conaghan PG, Ulff-Moller Dahl L, Terslev L, Altman RD, Becce F, Ginnerup-Nielsen E, Jensen L, Boesen M, Christensen R, Dal U, Bliddal H. Colchicine twice a day for hand osteoarthritis (COLOR): a double-blind, randomised, placebo-controlled trial. Lancet Rheumatol. 2023 May;5(5):e254-e262. doi: 10.1016/S2665-9913(23)00065-6. Epub 2023 Apr 4. PMID 38251589

DOCUMENTS (1):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04601883/Prot_000.pdf